CLINICAL TRIAL: NCT01170962
Title: A Phase 2B Study of BMS-790052 in Combination With Peginterferon Alfa-2a and Ribavirin in Chronic Hepatitis C Genotype 1 Infected Subjects Who Are Null or Partial Responders to Prior Treatment With Peginterferon Alfa Plus Ribavirin Therapy
Brief Title: Study of the Anti-HCV Drug (BMS-790052) Combined With Peginterferon and Ribavirin in Patients Who Failed Prior Treatment
Acronym: HEPCAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI444-011; 2010-019378-34 (EudraCT Number)
Record Dates: First submitted 2010-07-16; First posted 2010-07-28 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1: BMS-790052 plus peginterferon alfa-2a and ribavirin (Experimental): (prior null responders)
  Interventions: Drug: BMS-790052; Drug: peginterferon alfa-2a; Drug: ribavirin
- Arm 2: BMS-790052 plus peginterferon alfa-2a and ribavirin (Experimental): (prior null responders)
  Interventions: Drug: BMS-790052; Drug: peginterferon alfa-2a; Drug: ribavirin
- Arm 3: BMS-790052 plus peginterferon alfa-2a and ribavirin (Experimental): (prior partial responders)
  Interventions: Drug: BMS-790052; Drug: peginterferon alfa-2a; Drug: ribavirin
- Arm 4: BMS-790052 plus peginterferon alfa-2a and ribavirin (Experimental): (prior partial responders)
  Interventions: Drug: BMS-790052; Drug: peginterferon alfa-2a; Drug: ribavirin
- Arm 5: Placebo plus peginterferon alfa-2a and ribavirin (Experimental): (prior partial responders only)
  Interventions: Drug: Placebo; Drug: peginterferon alfa-2a; Drug: ribavirin

INTERVENTIONS:
Drug: BMS-790052 — Film coated tablet, Oral, 20 mg, once daily, 24 weeks
  Arms: Arm 1: BMS-790052 plus peginterferon alfa-2a and ribavirin; Arm 3: BMS-790052 plus peginterferon alfa-2a and ribavirin
Drug: BMS-790052 — Film coated Tablet, Oral, 60 mg, once daily (divided dose taken BID), 48 weeks
  Arms: Arm 2: BMS-790052 plus peginterferon alfa-2a and ribavirin; Arm 4: BMS-790052 plus peginterferon alfa-2a and ribavirin
Drug: Placebo — Film coated tablet, Oral, 0mg, Once daily, 24 weeks
  Arms: Arm 5: Placebo plus peginterferon alfa-2a and ribavirin
Drug: peginterferon alfa-2a — Solution for injection, Subcutaneous injection, 180 µg, weekly, 24 or 48 weeks
  Other Names: Pegasys®
Drug: ribavirin — Film coated tablet, Oral, 1,000 or 1,200 mg based on weight, divided dose taken twice a day (BID), 48 weeks
  Other Names: Copegus®

SUMMARY:
The purpose of this study is to determine whether BMS-790052 added to Peginterferon Alfa-2a and ribavirin can result in higher cure rates in patients who previously failed therapy and may have limited response to retreatment with Peginterferon Alfa-2a and ribavirin alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects chronically infected with HCV genotype 1
* Non-responder to prior therapy with peginterferon alfa and ribavirin
* HCV RNA viral load of 100,00 IU/mL
* Results of a liver biopsy ≤ 24 months prior to randomization consistent with chronic HCV infection; for compensated cirrhotics can be any time prior to randomization (compensated cirrhotics biopsy enrollment will be capped at 25% of randomized study population)
* Ultrasound, CT scan or MRI results 12 months prior to randomization that do not demonstrate hepatocellular carcinoma
* Body Mass Index (BMI) of 18 to 35 kg/m2

Exclusion Criteria:

* Positive for Hepatitis B infection (HBsAg) or HIV-1/HIV-2 antibody at screening
* Evidence of medical condition associated with chronic liver disease other than HCV
* Evidence of decompensated cirrhosis based on radiologic criteria or biopsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (69):
- United States (35):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - Scripps Clinic, La Jolla, California
  - CLI, Los Angeles, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - University Of California At San Francisco, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Transplant Center And Hepatology Clinic, B-154, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - University Of Florida Hepatology, Gainesville, Florida
  - Miami Research Associates, South Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Johns Hopkins Medical Institutions, Lutherville, Maryland
  - The Research Institute, Springfield, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Samuel S. Stratton Vamc, Albany, New York
  - James Sungsik Park, M.D. C.N.S.C., Great Neck, New York
  - Upper Delaware Valley Infectious Diseases, Pc, Monticello, New York
  - University Of Rochester Medical Center, Rochester, New York
  - James J Peters Vamc, The Bronx, New York
  - University Of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Nashville Medical Research Institute, Nashville, Tennessee
  - North Texas Research Institute, Arlington, Texas
  - Liver Associates Of Texas, Houston, Texas
  - St. Luke'S Episcopal Hospital - Baylor College Of Medicine, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Dean Clinic, Madison, Wisconsin
- Argentina (2):
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- Australia (6):
  - Local Institution, Randwick, New South Wales
  - Local Institution, Clayton, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Prahan, Victoria
  - Local Institution, Fremantle, Western Australia
  - Local Institution, Perth, Western Australia
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Toronto, Ontario
- Denmark (3):
  - Local Institution, Aarhus
  - Local Institution, Hvidovre
  - Local Institution, Odense
- France (6):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Lyon
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (4):
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
  - Local Institution, Hanover
- Italy (2):
  - Local Institution, Cisanello (pisa)
  - Local Institution, Pavia
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
- Puerto Rico (2):
  - Instituto De Investigacion Cientifica Del Sur, Ponce
  - Local Institution, San Juan
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 69 sites in 11 countries.
Pre-assignment Details: A total of 512 participants were enrolled and 421 participants were randomized (2 randomized participants were not treated: 1 due to positive pregnancy test and 1 no longer met criteria). Remaining 91 participants were not randomized as; 73 no longer met study criteria, 15 withdrew consent, 1 due to administrative reason and 2 for other reasons.
Groups:
- Daclatasvir (20 mg): Prior Null and Partial Responders: Participants (prior null or partial responders) received daclatasvir tablets 20 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Daclatasvir (60 mg): Prior Null and Partial Responders: Participants (prior null or partial responders) received daclatasvir tablets 60 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Placebo: Partial Responders: Participants who were prior partial responders received placebo matched with daclatasvir tablets orally, once daily for 24 weeks. Participants received pegIFNα-2a 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for 48 weeks and followed post treatment for 24 weeks. Prior partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
Period: Treatment Period
Arm/Group | Daclatasvir (20 mg): Prior Null and Partial Responders | Daclatasvir (60 mg): Prior Null and Partial Responders | Placebo: Partial Responders
Started | 203 | 199 | 17
No PDR | 145 | 127 | 17
PDR -Randomized to 24 Weeks pegIFNα--2a | 30 | 36 | 0
PDR -Randomized to 48 Weeks Follow--up | 28 | 36 | 0
Completed | 76 | 88 | 5
Not Completed | 127 | 111 | 12
Not completed — Lack of Efficacy | 96 | 91 | 7
Not completed — Adverse Event | 11 | 12 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Participant no longer meets criteria | 0 | 1 | 0
Not completed — Request to discontinue treatment | 7 | 3 | 1
Not completed — Completed 24 Week treatment period only | 10 | 2 | 0
Period: Follow up Period
Arm/Group | Daclatasvir (20 mg): Prior Null and Partial Responders | Daclatasvir (60 mg): Prior Null and Partial Responders | Placebo: Partial Responders
Started | 198 (Out of 203 participants who entered the treatment period, 198 continued in the follow-up period.) | 192 (Out of 199 participants who entered the treatment period, 192 continued in the follow-up period.) | 15 (Out of 17 participants who entered the treatment period, 15 continued in the follow-up period.)
Completed | 159 | 165 | 9
Not Completed | 39 | 27 | 6
Not completed — Withdrawal by Subject | 14 | 10 | 2
Not completed — Lost to Follow-up | 13 | 8 | 1
Not completed — Death | 2 | 2 | 0
Not completed — Others | 10 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Daclastavir (20mg): Prior Null and Partial Responders: Participants (prior null or partial responders) received daclatasvir tablets 60 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Daclastavir (60mg): Prior Null and Partial Responders: Participants (prior null or partial responders) received daclatasvir tablets 20 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Placebo: Prior Partial Responders: Participants who were prior partial responders received placebo matched with daclatasvir tablets orally, once daily for 24 weeks. Participants received pegIFNα-2a 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for 48 weeks and followed post treatment for 24 weeks. Prior partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Total: Total of all reporting groups
Arm/Group | Daclastavir (20mg): Prior Null and Partial Responders | Daclastavir (60mg): Prior Null and Partial Responders | Placebo: Prior Partial Responders | Total
Number analyzed (Participants) | 203 | 199 | 17 | 419
Age, Customized [Number; unit: participants]
  21-65 years | 192 | 189 | 15 | 396
  >=65 years | 11 | 10 | 2 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 72 | 4 | 146
  Male | 133 | 127 | 13 | 273

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as undetectable Hepatitis C virus RNA at both Weeks 4 and 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 4, Week 12
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir (20 mg): Prior Null Responders; Daclatasvir (20 mg): Prior Partial Responders; Daclatasvir (60 mg): Prior Partial Responders: Participants received daclatasvir tablets 20 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Daclatasvir (60 mg): Prior Null Responders: Participants received daclatasvir tablets 60 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 133 | 132 | 70 | 67 | 17
percentage of participants | 18.0 [13.8 to 22.3] | 19.7 [15.3 to 24.1] | 25.7 [19.0 to 32.4] | 35.8 [28.3 to 43.3] | 0 [0.0 to 0.0]

2. Primary Outcome: Percentage of Participants With 24-week Sustained Virologic Response (SVR24)
Description: SVR24 was defined as undetectable RNA (Hepatitis C Virus [HCV] RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at follow-up Week 24. TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Follow-up Week 24
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir (60 mg): Prior Partial Responders: Participants received daclatasvir tablets 60 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 133 | 132 | 70 | 67 | 17
percentage of participants | 18.8 [14.5 to 23.1] | 22.0 [17.4 to 26.6] | 24.3 [17.7 to 30.9] | 43.3 [35.5 to 51.0] | 0 [0.0 to 0.0]

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs) and Who Died On-treatment
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity; or was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From first dose to last dose plus 7 days, up to 49 weeks
Population: Safety population included all treated participants.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (20 mg): Prior Null and Partial Responders | Daclatasvir (60 mg): Prior Null and Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 203 | 199 | 17
participants
  SAEs | 14 | 11 | 3
  AEs Leading to Discontinuation of Treatment | 11 | 12 | 3
  Death | 0 | 0 | 1

4. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as undetectable RNA ie., Hepatitis C virus (HCV) RNA <lower limit of quantitation [LLOQ], target not detected (TND) at Week 4. TND was 10 IU/mL. HCV RNA levels were measured by the Roche Cobas® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 4
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir (60 mg): Prior Null Responders: Participants (prior null or partial responders) received daclatasvir tablets 60 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Placebo: Prior Partial Responders: Participants who were prior partial responders received placebo matched with daclatasvir tablets orally, once daily along with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily up to 24 weeks. Participants continued to receive pegIFNα-2a and ribavirin, up to 48 weeks followed by a post treatment follow-up period of 24 weeks. Prior partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 133 | 132 | 70 | 67 | 17
percentage of participants | 21.8 [17.2 to 26.4] | 21.2 [16.7 to 25.8] | 25.7 [19.0 to 32.4] | 38.8 [31.2 to 46.4] | 0 [0.0 to 0.0]

5. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as undetectable RNA ie., Hepatitis C virus (HCV) RNA <lower limit of quantitation [LLOQ], target not detected (TND) at Week 12. TND was 10 IU/mL. HCV RNA levels were measured by the Roche Cobas® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 133 | 132 | 70 | 67 | 17
percentage of participants | 30.1 [25.0 to 35.2] | 34.1 [28.8 to 39.4] | 44.3 [36.7 to 51.9] | 56.7 [49.0 to 64.5] | 0 [0.0 to 0.0]

6. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Week 12 (SVR12)
Description: SVR12 was defined as undetectable RNA ie., Hepatitis C virus (HCV) RNA <lower limit of quantitation (LLOQ), target not detected (TND) at follow-up Week 12. TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Follow-up Week 12
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 133 | 132 | 70 | 67 | 17
percentage of participants | 19.5 [15.1 to 24.0] | 23.5 [18.8 to 28.2] | 25.7 [19.0 to 32.4] | 47.8 [39.9 to 55.6] | 0 [0.0 to 0.0]

7. Secondary Outcome: Number of Participants With Genotypic-1A Substitution at Baseline, On-treatment and During Follow-up Associated With Virologic Failures
Description: Non-structural protein 5A of HCV resistance associated polymorphism in GT-1a samples included M28L/T/V, Q30H, L31M, H54Y, H58C/D/N/P/Q, E62D and Y93C.
Time Frame: Baseline to follow-up Week 48
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Groups:
- Daclatasvir (60 mg): Prior Partial Responders: Participants who were prior partial responders received placebo matched with daclatasvir tablets orally, once daily for 24 weeks. Participants received pegIFNα-2a 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for 48 weeks and followed post treatment for 24 weeks. Prior partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy.
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders
Number analyzed (Participants) | 83 | 86 | 50 | 37
participants
  M28: L/T/V: Baseline (n=78,84,49,36) | 2 | 3 | 1 | 3
  M28: L/T/V: On-Treatment (n= 60,57,34,22) | 2 | 3 | 1 | 2
  M28: L/T/V: Relapsers (n=10,12,7,3) | 0 | 0 | 0 | 0
  Q30: H: Baseline (n=78,0,0,36) | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 1
  Q30: H: On-Treatment (n= 60,0,0,22) | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 0
  Q30: H:Relapsers (n=10,0,0,3) | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 0
  L31: M: Baseline (n=78,84,49,36) | 5 | 1 | 1 | 2
  L31: M: On-Treatment (n= 60,57,34,22) | 5 | 1 | 0 | 2
  L31: M: Relapsers (n=10,12,7,3) | 0 | 0 | 1 | 0
  H54: Y: Baseline (n=0,84,49,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 2 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  H54: Y: On-Treatment (n=0,57,34,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 2 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  H54: Y: Relapsers (n=0,12,7,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 0 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  H58: C/D/N/P/Q: Baseline (n=78,84,49,0) | 4 | 3 | 3 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  H58: C/D/N/P/Q: On-Treatment (n= 60,57,34,0) | 4 | 3 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  H58: C/D/N/P/Q: Relapsers (n=10,12,7,3) | 0 | 0 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  E62: D: Baseline (n=78,84,49,0) | 1 | 3 | 2 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  E62: D: On-Treatment (n= 60,57,34,0) | 1 | 2 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  E62: D: Relapsers (n=10,12,7,0) | 0 | 1 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  Y93: C: Baseline (n=0,84,49,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 1 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  Y93: C: On-Treatment (n= 0,57,34,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 1 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  Y93: C: Relapsers (n=0,12,7,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 0 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.

8. Secondary Outcome: Number of Participants With Genotypic-1B Substitution at Baseline, On-treatment and During Follow-up Associated With Virologic Failures
Description: Non-structural protein 5A of HCV resistance associated polymorphisms in GT-1b samples, included L28M/V, R30H/Q, L31M, Q54H/N/Y, P58A/Q/S, Q62E/K/N/R/S, A92T/V and Y93F/H.
Time Frame: Baseline to follow-up Week 48
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (20 mg): Prior Null Responders | Daclatasvir (60 mg): Prior Null Responders | Daclatasvir (20 mg): Prior Partial Responders | Daclatasvir (60 mg): Prior Partial Responders
Number analyzed (Participants) | 44 | 38 | 20 | 29
participants
  L28: M/V: Baseline (n=43,37,19,0) | 1 | 1 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  L28: M/V: On-Treatment (n=19,20,6,0) | 1 | 1 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  L28: M/V: Relapsers (n=7,6,2,0) | 0 | 0 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  R30: H/Q: Baseline (n=43,37,19,27) | 4 | 5 | 1 | 1
  R30: H/Q: On-Treatment (n=19,20,6,5) | 4 | 3 | 0 | 0
  R30: H/Q: Relapsers (n=7,6,2,9) | 0 | 2 | 1 | 1
  L31: M: Baseline (n=43,37,19,27) | 4 | 5 | 1 | 1
  L31: M: On-Treatment (n=19,20,6,5) | 2 | 4 | 0 | 0
  L31: M: Relapsers (n=7,6,2,9) | 1 | 0 | 1 | 1
  Q54: H/N/Y: Baseline (n=43,37,19,27) | 18 | 20 | 9 | 8
  Q54: H/N/Y: On-Treatment (n=19,20,6,5) | 9 | 12 | 5 | 2
  Q54: H/N/Y: Relapsers (n=7,6,2,9) | 5 | 1 | 0 | 2
  P58: A/Q/S: Baseline (n=43,37,19,27) | 3 | 7 | 2 | 3
  P58: A/Q/S: On-Treatment (n=19,20,6,5) | 2 | 3 | 1 | 0
  P58: A/Q/S: Relapsers (n=7,6,2,9) | 0 | 2 | 0 | 1
  Q62: E/K/N/R/S: Baseline (n=43,37,19,27) | 5 | 1 | 2 | 1
  Q62: E/K/N/R/S: On-Treatment (n=19,20,6,5) | 3 | 1 | 1 | 0
  Q62: E/K/N/R/S: Relapsers (n=7,6,2,9) | 0 | 0 | 0 | 1
  A92: T/V: Baseline (n=43,37,19,0) | 2 | 3 | 3 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  A92: T/V: On-Treatment (n=0,20,6,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 2 | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  A92: T/V: Relapsers (n=0,6,2,0) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 0 | 0 | NA — Data was not analyzed as no participant was evaluable at the specified time-point.
  Y93: F/H: Baseline (n=43,37,0,27) | 1 | 5 | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 3
  Y93: F/H: On-Treatment (n=0,20,0,5) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 4 | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 0
  Y93: F/H: Relapsers (n=0,6,0,9) | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 1 | NA — Data was not analyzed as no participant was evaluable at the specified time-point. | 2

9. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Who Died During Follow-up Period
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From day 8 post last dose of treatment up-to Week 72
Population: Safety population included all treated participants.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (20 mg): Prior Null and Partial Responders | Daclatasvir (60 mg): Prior Null and Partial Responders | Placebo: Prior Partial Responders
Number analyzed (Participants) | 198 | 192 | 15
participants
  SAEs | 6 | 7 | 0
  Death | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 7 days, up to 49 weeks
Description: On-Treatment Period
Groups:
- Daclatasvir (20 mg): Prior Null and Partial Responders: Participant (prior null or partial responders) received daclatasvir tablets 20 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
- Daclatasvir (60 mg): Prior Null and Partial Responders: Participant (prior null or partial responders) received daclatasvir tablets 60 mg orally once daily, pegylated-interferon alfa-2a (pegIFNα-2a) injection 180 µg/0.5 mL subcutaneously once weekly, ribavirin tablets 1000-1200 mg orally twice daily for 24 weeks. At Week 24, participants with a protocol defined response (PDR: HCV RNA <LOQ at Week 4, undetectable HCV RNA at Week 12) were randomized (1:1) to either a follow-up period of 48 weeks or received pegIFNα-2a and ribavirin for 24 weeks and then followed for 24 weeks. Participants with no PDR continued to receive pegIFNα-2a and ribavirin, for an additional 24 weeks and followed up for 24 weeks. Prior null responders: <1 log10 HCV RNA decrease from baseline at or after 4 weeks, or <2 log10 decrease from baseline in HCV RNA at or after Week 12 of IFN-based therapy. Prior Partial responders: >2 log10 decrease in HCV RNA from baseline at Week 12 of IFN-based therapy but detectable HCV RNA when therapy was discontinued.
Arm/Group | Daclatasvir (20 mg): Prior Null and Partial Responders | Daclatasvir (60 mg): Prior Null and Partial Responders | Placebo: Prior Partial Responders
Serious Adverse Events (participants affected / at risk) | 14/203 | 11/199 | 3/17
Other Adverse Events (participants affected / at risk) | 190/203 | 195/199 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir (20 mg): Prior Null and Partial Responders (N=203) | Daclatasvir (60 mg): Prior Null and Partial Responders (N=199) | Placebo: Prior Partial Responders (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Bladder perforation (Renal and urinary disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cat scratch disease (Infections and infestations) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 1 | 0
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Retinal exudates (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir (20 mg): Prior Null and Partial Responders (N=203) | Daclatasvir (60 mg): Prior Null and Partial Responders (N=199) | Placebo: Prior Partial Responders (N=17)
Anaemia (Blood and lymphatic system disorders) | 43 | 28 | 4
Anxiety (Psychiatric disorders) | 13 | 16 | 1
Asthenia (General disorders) | 55 | 38 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 47 | 3
Decreased appetite (Metabolism and nutrition disorders) | 38 | 36 | 4
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 7 | 10 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 7 | 3
Gingival abscess (Infections and infestations) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 8 | 5 | 1
Nasopharyngitis (Infections and infestations) | 7 | 10 | 1
Photophobia (Eye disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 38 | 38 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 10 | 2
Vomiting (Gastrointestinal disorders) | 19 | 16 | 2
Amnesia (Nervous system disorders) | 4 | 3 | 1
Blepharitis (Eye disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 22 | 11 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Injection site erythema (General disorders) | 15 | 14 | 0
Injection site haematoma (General disorders) | 0 | 3 | 1
Pain (General disorders) | 9 | 9 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 14 | 2
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 31 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 39 | 65 | 4
Feeling abnormal (General disorders) | 3 | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 33 | 4
Nausea (Gastrointestinal disorders) | 55 | 45 | 3
Neutropenia (Blood and lymphatic system disorders) | 31 | 31 | 4
Palpitations (Cardiac disorders) | 3 | 2 | 1
Pharyngitis (Infections and infestations) | 3 | 2 | 1
Sleep disorder (Psychiatric disorders) | 12 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 19 | 12 | 3
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 7 | 10 | 2
Dyspepsia (Gastrointestinal disorders) | 13 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 39 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 6 | 4 | 1
Insomnia (Psychiatric disorders) | 53 | 53 | 5
Oedema peripheral (General disorders) | 2 | 5 | 2
Urinary tract infection (Infections and infestations) | 9 | 5 | 1
Affect lability (Psychiatric disorders) | 4 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 36 | 42 | 1
Bronchitis (Infections and infestations) | 11 | 4 | 0
Constipation (Gastrointestinal disorders) | 11 | 5 | 1
Dry mouth (Gastrointestinal disorders) | 9 | 14 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 2
Weight decreased (Investigations) | 13 | 6 | 2
Cheilitis (Gastrointestinal disorders) | 5 | 3 | 1
Chills (General disorders) | 16 | 27 | 4
Depressed mood (Psychiatric disorders) | 4 | 1 | 1
Depression (Psychiatric disorders) | 25 | 23 | 3
Diarrhoea (Gastrointestinal disorders) | 26 | 32 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 15 | 2
Feeling hot (General disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 5 | 0
Influenza like illness (General disorders) | 55 | 59 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 9 | 2 | 2
Mucosal dryness (General disorders) | 3 | 2 | 1
Ocular hyperaemia (Eye disorders) | 2 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 55 | 63 | 3
Tachycardia (Cardiac disorders) | 6 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 14 | 0
Crying (General disorders) | 1 | 0 | 1
Eyelid disorder (Eye disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 4 | 3 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 5 | 6 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hypotension (Vascular disorders) | 3 | 1 | 1
Irritability (General disorders) | 29 | 42 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 1
Vertigo (Ear and labyrinth disorders) | 10 | 11 | 0
Cataract (Eye disorders) | 0 | 1 | 1
Drug dependence (Psychiatric disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 10 | 12 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Fatigue (General disorders) | 81 | 91 | 10
Headache (Nervous system disorders) | 71 | 63 | 7
Injection site rash (General disorders) | 3 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 19 | 2
Pollakiuria (Renal and urinary disorders) | 5 | 5 | 1
Pyrexia (General disorders) | 19 | 23 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.